CLINICAL TRIAL: NCT03594279
Title: Evaluation of a Community Engagement and Demand Creation Strategy for Childhood Diarrhea and Pneumonia in Pakistan
Brief Title: Community Mobilization and Incentivization for Childhood Diarrhea and Pneumonia
Acronym: CoMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Jai Kumar Das, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4676-WCH-ERC-17
Record Dates: First submitted 2018-06-28; First posted 2018-07-20 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Childhood Diarrhea; Childhood Pneumonia; Community Mobilisation; Sanitation and Hygiene; Community Incentives

STUDY DESIGN:
Intervention Model Description: The intervention is based on the Behavior Change Theory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community Mobilization (Experimental): This arm will receive specific messages regarding the prevention and management of childhood diarrhea and pneumonia. The investigators will form village committees (VC) consisting of prominent members of the community (6-8 in a group) to carry out awareness and motivational activities for the uptake of the identified interventions.
  Interventions: Behavioral: Community Mobilization; Behavioral: Community Mobilization and Community Incentive
- Community Mobilization and Community Incentive (Experimental): In this arm, along with the interventions in the community mobilization arm, community based incentives will also be provided. The clusters which improve the practices for preventive and curative strategies for diarrhea and pneumonia will receive community-based incentive including structural benefits linked to health including tube wells, water supply, toilets in community/schools, water storage facility or any other incentive as decided with the respective village committees.
  Interventions: Behavioral: Community Mobilization and Community Incentive
- Control (No Intervention): This arm will receive the routine standard of care.

INTERVENTIONS:
Behavioral: Community Mobilization — Community Mobilization
  Arms: Community Mobilization
Behavioral: Community Mobilization and Community Incentive — Community Mobilization and Community Incentive
  Arms: Community Mobilization; Community Mobilization and Community Incentive

SUMMARY:
Childhood diarrhea and pneumonia remains the leading cause of mortality among children under five years of age in Pakistan. The prevalence of diarrhea in Pakistan has increased from 15% in 1990 to 23% in 2013 while there has been no progress in the prevalence of pneumonia and it has been almost constant over the last two decades. The coverage of preventive and therapeutic interventions for childhood diarrhea and pneumonia also remains low. This study aims to improve the adherence to recommended preventive and curative practices for childhood diarrhea and pneumonia.

DETAILED DESCRIPTION:
Study Components and Objectives:

This study will be conducted in two phases:

1. Formative phase: The objective of this phase is to assess the existing care seeking practices and care provision for childhood diarrhea and pneumonia and identify the existing barriers and facilitators for care seeking for childhood diarrhea and pneumonia.
2. Cluster Randomized Trial: (CoMIC Trial - Community Mobilization and Community Incentivization): The objective of this phase is to assess the impact of a community engagement and demand creation strategy involving an community-based incentive scheme on adherence to recommended preventive and curative practices for diarrhea and pneumonia among children under five years of age.

Study site: This study will be conducted in Tando Muhammad Khan, which is a rural district in the province of Sindh. This would a three and half year study with two year of intervention period.

Study design: This study will follow a mixed methodology approach with a formative research component followed by a prospective two arm cluster randomized controlled trial (cRCT).

Formative Phase: The following activities will be conducted in the formative phase:

* GIS Mapping: for the whole district to map all the government health facilities, schools, major religious places (mosques), water supply sources and roads.
* Qualitative research: comprising of focus group discussion (FGDs) and in-depth interviews (IDIs) with all stakeholders. These would also identify the potential non-cash incentives that the community wants and could be attractive
* Baseline Household Survey: Baseline survey will be conducted at the household level and will gather information on health care practices pertaining to childhood diarrhea and pneumonia, immunization, socio-economic indicators, childhood nutrition indicators and WASH indicators. LHWs working in the study area and their geographic spread will also be identified.

Randomized Controlled Trial:

-Randomization: After the mapping and formative research, the clusters (villages) will be randomly allocated to two intervention arms and a control arm by an independent statistician in the ratio of 1:1:1.

Sample size: The sample size was calculated with a power of 0.8 and alpha of 0.05 giving 14 clusters per arm (maximum sample size). These clusters will be randomly allocated to three arms.

Intervention:

Arm 1: In Arm 1, separate male and female village committees (VC) consisting of prominent members of the community including local elites/leaders (6 to 8 in a group) in all the villages will be formed and they would be trained on specific messages regarding the prevention and management of childhood diarrhea and pneumonia. The VCs would carry out awareness and motivational activities for the uptake of the identified interventions. They would also facilitate two hour group meetings to be held twice every month in every village of their catchment area and focus on issues pertaining to childhood nutrition, WASH, vaccines and management of diarrhea and pneumonia in children. Apart from these, there would researcher led awareness sessions in this intervention cluster and specific sessions for children would also be conducted. These sessions would focus on providing education and encourage community participation. Group activities would also identify community level health, nutrition and sanitation problems, and to find locally feasible strategies to address them.

Arm 2: In the second intervention cluster; in addition to the interventions in Arm 1, the areas which improve the practices for preventive and curative strategies for diarrhea and pneumonia will receive community-based incentive. This would be a unique incentive scheme as all the previous financial incentive programs whether conditional or unconditional cash transfers, voucher schemes, social insurance schemes have targeted individuals and all these incentives were based on improving individual practices. The financial incentive proposed is unique as this initiative which would benefit the community as a whole and incentives based on improvement in the composite coverage of three indicators:

* Age-appropriate immunization 12-23 months
* ORS use for diarrhea
* Sanitation index (which is a score based on personal, household and environmental hygiene) The incentives would include structural benefits linked to health including tube wells, water supply, toilets in community/schools, water storage facility or any other incentive as decided with the respective village committees. The total cost of these incentives would be shared by the project (75%) and the community (25%), to improve ownership. The contribution from the community could also be in-kind including labor etc.

Arm 3: This arm will receive routine standard of care.

ELIGIBILITY:
Inclusion Criteria:

* People residing in the villages in the selected study site and consent to participate.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Age-appropriate immunization 12-23 months | At six months of intervention
ORS use for diarrhea | At six months of intervention
Mean Sanitation Index | At six months of intervention
  The scale is focused on 12 components. All the components are valued equally and can be scored '0' (for 'No') or '1' (for 'Yes'). These would be summed up for each household for a total possible score of 12 and a range of 0-12. Higher score represents a better outcome. It comprises of the following three subscales:
  1. Drinking water - possible score of minimum 0 and maximum 3
     * Interior water storage container is covered;
     * Exterior water storage container is cleaned;
     * Water present in water storage container
  2. Food - possible score of minimum 0 and maximum 3
     * Clean dishes are covered;
     * Clean dishes are kept high;
     * All food is covered
  3. Domestic hygiene - possible score of minimum 0 and maximum 6
     * No trash outside the house;
     * No trash inside the house;
     * No unrestrained animals in patio or house;
     * No accumulation of dirty clothes;
     * Insignificant number of flies in house;
     * No standing water in patio or around house
Age-appropriate immunization 12-23 months | At 12 months of intervention
ORS use for diarrhea | At 12 months of intervention
Mean Sanitation Index | At 12 months of intervention
  The scale is focused on 12 components. All the components are valued equally and can be scored '0' (for 'No') or '1' (for 'Yes'). These would be summed up for each household for a total possible score of 12 and a range of 0-12. Higher score represents a better outcome. It comprises of the following three subscales:
  1. Drinking water - possible score of minimum 0 and maximum 3
     * Interior water storage container is covered;
     * Exterior water storage container is cleaned;
     * Water present in water storage container
  2. Food - possible score of minimum 0 and maximum 3
     * Clean dishes are covered;
     * Clean dishes are kept high;
     * All food is covered
  3. Domestic hygiene - possible score of minimum 0 and maximum 6
     * No trash outside the house;
     * No trash inside the house;
     * No unrestrained animals in patio or house;
     * No accumulation of dirty clothes;
     * Insignificant number of flies in house;
     * No standing water in patio or around house
Age-appropriate immunization 12-23 months | At 24 months of intervention
ORS use for diarrhea | At 24 months of intervention
Mean Sanitation Index | At 24 months of intervention
  The scale is focused on 12 components. All the components are valued equally and can be scored '0' (for 'No') or '1' (for 'Yes'). These would be summed up for each household for a total possible score of 12 and a range of 0-12. Higher score represents a better outcome. It comprises of the following three subscales:
  1. Drinking water - possible score of minimum 0 and maximum 3
     * Interior water storage container is covered;
     * Exterior water storage container is cleaned;
     * Water present in water storage container
  2. Food - possible score of minimum 0 and maximum 3
     * Clean dishes are covered;
     * Clean dishes are kept high;
     * All food is covered
  3. Domestic hygiene - possible score of minimum 0 and maximum 6
     * No trash outside the house;
     * No trash inside the house;
     * No unrestrained animals in patio or house;
     * No accumulation of dirty clothes;
     * Insignificant number of flies in house;
     * No standing water in patio or around house

SECONDARY OUTCOMES:
Handwashing with soap at important time | At 24 months of intervention
Exclusive breastfeeding rates - children who are exclusively breastfed at 6 months of age | At 24 months of intervention
Care seeking for severe cases of childhood diarrhea and pneumonia - parents/caregivers who sought care for child with diarrhea/pneumonia | At 24 months of intervention
Prevalence of Diarrhea and pneumonia | At 24 months of intervention
Open defecation rates | At 24 months of intervention
Total cost (unit cost and cost effectiveness) | At 24 months of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Das JK, Salam RA, Padhani ZA, Rizvi A, Mirani M, Jamali MK, Chauhadry IA, Sheikh I, Khatoon S, Muhammad K, Bux R, Naqvi A, Shaheen F, Ali R, Muhammad S, Cousens S, Bhutta ZA. An innovative Community Mobilisation and Community Incentivisation for child health in rural Pakistan (CoMIC): a cluster-randomised, controlled trial. Lancet Glob Health. 2025 Jan;13(1):e121-e133. doi: 10.1016/S2214-109X(24)00428-5. PMID 39706650
- [Derived] Das JK, Siddiqui F, Padhani ZA, Khan MH, Jabeen S, Mirani M, Mughal S, Baloch S, Sheikh I, Khatoon S, Muhammad K, Gangwani M, Nathani K, Salam RA, Bhutta ZA. Health behaviors and care seeking practices for childhood diarrhea and pneumonia in a rural district of Pakistan: A qualitative study. PLoS One. 2023 May 16;18(5):e0285868. doi: 10.1371/journal.pone.0285868. eCollection 2023. PMID 37192190